CLINICAL TRIAL: NCT03791112
Title: A Phase I Study of BPI-16350 in Patients with Advanced Solid Tumor
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTP-66711
Record Dates: First submitted 2018-12-29; First posted 2019-01-02 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Advanced Solid Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- 50mg QD (Experimental): Participants received 50 mg BPI-16350 administered orally (PO), once daily (QD), in a fasted state on Days 1 to 28 of a 28-day cycle.
  Interventions: Drug: BPI-16350
- 100mg QD (Experimental): Participants received 100 mg BPI-16350 administered orally (PO), once daily (QD), in a fasted state on Days 1 to 28 of a 28-day cycle.
  Interventions: Drug: BPI-16350
- 200mg QD (Experimental): Participants received 200 mg BPI-16350 administered orally (PO), once daily (QD), in a fasted state on Days 1 to 28 of a 28-day cycle.
  Interventions: Drug: BPI-16350
- 300mg QD (Experimental): Participants received 300 mg BPI-16350 administered orally (PO), once daily (QD), in a fasted state on Days 1 to 28 of a 28-day cycle.
  Interventions: Drug: BPI-16350
- 400mg QD (Experimental): Participants received 400 mg BPI-16350 administered orally (PO), once daily (QD), in a fasted state on Days 1 to 28 of a 28-day cycle.
  Interventions: Drug: BPI-16350
- 500mg QD (Experimental): Participants received 500 mg BPI-16350 administered orally (PO), once daily (QD), in a fasted state on Days 1 to 28 of a 28-day cycle.
  Interventions: Drug: BPI-16350

INTERVENTIONS:
Drug: BPI-16350 — BPI-16350 capsules administered orally

SUMMARY:
This was an open-label Phase I study. The primary objective of the study was to assess safety, tolerability, efficacy, and pharmacokinetic characteristics of BPI-16350 in different dose groups.

DETAILED DESCRIPTION:
The study was divided into two sections: dose escalation section and expanded enrollment section.

In dose escalation section, BPI-16350 were administered orally once daily (QD) to patients with locally advanced or metastatic solid tumors in different dose levels.The study was designed to evaluate the safety, tolerability, and pharmacokinetics of single dose and multiple doses of BPI-16350.

In expanded enrollment section, based on the results of dose escalation section, BPI-16350 were administered orally to patients with locally advanced or metastatic solid tumors, to further evaluate the safety, tolerability, and pharmacokinetics of BPI-16350.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological diagnosis of patients with advanced solid tumors, pateints couldn't be benefit from the existing standard treatment options, and patients were not suitable for surgical resection or radiation therapy for the purpose of cure;
2. There were measurable lesions defined in RECIST v. 1.1. Tumor lesions that had previously received radiotherapy or other local treatment were considered as measurable lesions only when disease progression at the treatment site was clearly recorded after treatment;
3. Age ≥ 18 and ≤ 70 years old;
4. Expected survival ≥ 12 weeks;
5. Eastern Cancer Cooperative Group (ECOG) performance status 0-1;
6. Adequate bone marrow, hepatic, and renal function;
7. Patients of child bearing potential must agree to take contraception during the study and for 90 days after the last day of treatment;
8. All acute toxicity of previous anti-tumor treatment or surgery is relieved to baseline severity or NCI CTCAE version 4.03 ≤ 1 (except for hair loss or other toxicity that the investigator believes has no safety risk to the patient);
9. Voluntarily enroll and sign informed consent, follow the trial treatment plan and visit plan.

Exclusion Criteria:

1. Received other anti-tumor treatments (including chemotherapy, radiotherapy, immunotherapy and experimental treatment) within 28 days (for myelosuppressive drugs or treatment) or within 14 days (for non-myelosuppressive drugs or treatment) before receiving the study drug;
2. Previous treatments for other CDK4/6 inhibitors, such as Abemaciclib (VERZENIOTM, LY2835219), Palbociclib (IBRANCE®, PD0332991), Ribociclib (KISQALI®, LEE-011), Birosiclib (XZP-) 3287), SHR-6390, Trilaciclib and G1T-38, etc.;
3. Any of the following cardiac criteria: unexplained or cardiovascular causes of threatened syncope or syncope, ventricular tachycardia, ventricular fibrillation or cardiac arrest. Corrected QT interval prolongation [A mean corrected QT interval (male QTcF > 450 msec or female QTcF > 470 msec) obtained from 3 electrocardiogram (ECG) examinations at rest. Various clinically significant cardiac rhythm, conduction, resting ECG morphological abnormalities, such as complete left bundle branch block, III degree block, II degree block, PR interval > 250 msec;
4. Clinically active bacterial, fungal or viral infections (eg active hepatitis B (HBV), hepatitis C (HCV), human immunodeficiency virus (HIV) and syphilis positive, no other activities required at the time of enrollment Screening for sexual infections);
5. Patients who had undergone autologous or allogeneic organ or stem cell transplantation; patients who had undergone major surgery or severe trauma within 4 weeks prior to the first dose;
6. The patient received the following treatment within 7 days prior to entering the study: a known or potent CYP3A inhibitor or inducer, and a drug primarily metabolized by CYP2C19; or consumed grapefruit and grapefruit juice;
7. Patients who received anti-tumor treatment of Chinese herbal medicine within 1 week before the first dose;
8. There were primary CNS（central nervous system）malignant tumors. Patients with CNS metastases who failed local treatment. For patients with asymptomatic brain metastases, or stable clinical symptoms and no need for steroids and other treatments for brain metastases ≥ 28 days can be enrolled;
9. Have had other malignant tumors in the past 5 years, except for basal cell carcinoma and cervical carcinoma in situ after radical treatment;
10. Occurrence of venous/venous thrombosis within 6 months prior to the first dose, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism;
11. The prevalence of familial and/or acquired thrombophilia, such as the presence of genetic or acquired defects such as anticoagulant, coagulation factors, fibrinolytic proteins, or the presence of acquired risk factors with a high tendency to thromboembolism;
12. Any condition that affected the patient's swallowing of the drug, as well as conditions that seriously affect the absorption or pharmacokinetic parameters of the test drug, including uncontrollable nausea and vomiting, chronic gastrointestinal disease, gastrointestinal resection or surgical history;
13. It was known to be severely allergic to study drugs or any excipients;
14. The existence of drugs of abuse and patients whose medical, psychological or social conditions may interfere with or participate in the evaluation of the results of the study;
15. Any unstable systemic diseases (including active ≥CTCAE level 2 clinically serious infections, uncontrolled high blood pressure, unstable angina pectoris, congestive heart failure, severe liver and kidney or metabolic diseases, etc.);
16. Any condition that was unstable or may jeopardize patient safety and its compliance with the study;
17. Other conditions that the investigator believeed were not suitable for participation in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2019-07-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Participants with Adverse Events | 24 months
  The safety and tolerability variables include adverse events, physical examinations, vital signs , clinical laboratory evaluations including serum chemistry, hematology , and urinalysis, and electrocardiograms (ECGs) in triplicate,Incidence and nature of DLTs ( dose-limiting toxicity), To determine the MTD (maximum tolerated dose).

SECONDARY OUTCOMES:
Cmax | 1 month
  Day 1-7 for single dose, and day 1-28 for steady state
Half-life time | 1 month
  Day 1-7 for single dose, and day 1-28 for steady state
Tmax | Time to Cmax

OTHER OUTCOMES:
Progression-free survival | 6-24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Betta Pharmaceuticals Co., Hangzhou, Zhejiang Provice, China

IPD SHARING:
Plan to Share IPD: Undecided